CLINICAL TRIAL: NCT03647735
Title: Propofol Sedation in Orthopaedic Surgery Under Central Neuraxial Block: Patient-controlled Sedation Versus Target-controlled Infusion
Brief Title: Patient-controlled Sedation Versus Target-controlled Infusion in Orthopaedic Surgery Under Central Neuraxial Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FF-2017-265
Record Dates: First submitted 2018-08-01; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Patient-controlled Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PCS (Experimental): Patients in Group PCS (patient-controlled sedation) received intravenous (IV) propofol via a patient controlled analgesia (PCA) infusion pump. The machine was set to deliver a demand bolus dose of 0.25 mg/kg with 1-minute lockout interval, without basal infusion.The patient was instructed to press on a hand-held device as often as required, to achieve their desired level of comfort or sedation.
  Interventions: Other: patient-controlled sedation
- Group TCIS (Active Comparator): Patients in Group TCIS (target-controlled infusion sedation) received IV propofol via a target-controlled infusion (TCI) pump, targeted at an initial effect site concentration (Cet) of 0.6 μg/ml, using the Schnider pharmacokinetic model. Upon attainment of 0.6 μg/ml Cet, the patient's sedation level was assessed. The Cet was increased or reduced accordingly by 0.2 μg/ml to attain an OAA/S score of 3.
  Interventions: Other: patient-controlled sedation

INTERVENTIONS:
Other: patient-controlled sedation — Patient-controlled propofol boluses for patients undergoing elective orthopaedic surgery under central neuraxial block

SUMMARY:
Orthopaedic surgeries involving the legs can be done under nerve block, where patients will be numb of pain at the operated site but awake during surgery. Sedation can be given to allay anxiety and provide comfort throughout the surgery. Sedation can be given by the anaesthetic doctors by using target-comtrolled infusion pump, or self-administered by patients by means of specialised machines. This study compares two method of administration of sedation, patient-controlled sedation (PCS) versus target-controlled infusion sedation (TCIS) by anaesthetic doctors, in people undergoing orthopaedic surgeries under nerve block.

DETAILED DESCRIPTION:
Central neuraxial block (CNB) is one of the mainstays of anaesthesia methods in various disciplines particularly orthopaedic surgeries. However the state of consciousness can potentially cause patient anxiety thus sedation is often utilized as a mean to improve patient satisfaction and increase patient acceptance of CNB.

Conventionally, the anaesthesiologist administers sedatives for the patients. Propofol is the commonly used drug for sedation due to its favourable pharmacokinetic profile, which results in fast induction, easy control of depth of sedation and rapid recovery. It can be infused by using target-controlled infusion (TCI) devices where the anaesthetists titrates propofol by setting desired target plasma and effect site concentration. However it is difficult to judge precisely patient requirements for adequate patient sedation, comfort and analgesia as patients' needs differ.

Patient-controlled sedation (PCS) is a valid option, initially adapted from post surgery patient-controlled analgesia. It allows patients to titrate sedative medication to their comfort and therefore present an option that addresses the needs of patients with strong desire to maintain sense of control during procedures.

This study was designed to compare total propofol requirement between PCS versus TCI sedation (TCIS), complications and patient satisfaction, in patients undergoing lower limb orthopaedic surgery under CNB.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) I or II.
2. Aged 18-65 years.
3. Elective lower limb orthopaedic surgery under CNB anticipated to last for 1.5 to 2 hours

Exclusion Criteria:

1. Body Mass Index (BMI) > 30kg/m2
2. Unable to cooperate (eg. mental disorders, language barrier)
3. Drug abuse
4. Alcoholism (chronic daily alcohol intake greater than 75 g of pure alcohol for ≥ 2 years, where 75g of alcohol = 5 cans of beer, 1 bottle of wine or half a pint of distilled spirit)
5. Contraindications to the study drugs
6. Pregnancy
7. Significant pulmonary or cardiovascular diseases, including obstructive sleep apnoea and obesity hypoventilation syndrome
8. Features of difficult airway

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
total propofol requirement between PCS versus TCI sedation (TCIS) | Assessed from the beginning to the end of sedation, at the average of 120 minutes
  Total propofol requirement in both groups was calculated in mg/kg/hour.

SECONDARY OUTCOMES:
Patient satisfaction assessed by a 10-point numerical scale | Within one hour after recovery from sedation
  Assessed using a 10-point verbal numerical rating scale (1 to 10), where 1 was regarded as extremely dissatisfied and 10 extremely satisfied.
Complications including incidence of hypotension, bradycardia, hypopnea, oxygen desaturation and over sedation | Assessed from the beginning to the end of sedation, at the average of 120 minutes
  Documented as Yes or No for each specified complication

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Md Nor, MMED(Anaes), Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Wahlen BM, Kilian M, Schuster F, Muellenbach R, Roewer N, Kranke P. Patient-controlled versus continuous anesthesiologist-controlled sedation using propofol during regional anesthesia in orthopedic procedures--a pilot study. Expert Opin Pharmacother. 2008 Nov;9(16):2733-9. doi: 10.1517/14656566.9.16.2733. PMID 18937608
- [Result] Ekin A, Donmez F, Taspinar V, Dikmen B. Patient-controlled sedation in orthopedic surgery under regional anesthesia: a new approach in procedural sedation. Braz J Anesthesiol. 2013 Sep-Oct;63(5):410-4. doi: 10.1016/j.bjan.2012.07.012. PMID 24263045
- [Result] Singh T, Ravishankar M. Conscious sedation with propofol for surgeries under spinal anaesthesia: anaesthesiologist versus patient controlled. J Anaesthesiol Clin Pharmacol. 21:169-173, 2005.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03647735/Prot_SAP_000.pdf